CLINICAL TRIAL: NCT06260189
Title: Assessment Of Serum And Tissue Levels Of Cold-Inducible RNA-Binding Protein In Patients With Lichen Planus
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Elsayed, Aya Ahmed Elsayed, Sohag University
Other Study IDs: Soh-Med-24-01-02MD
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Assessment, Self
Keywords: Lichen Planus, Cold-inducible RNA-binding protein
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lichen Planus Cases: 40 cases with lichen planus from who skin biopsies and blood samples will be taken to assess cold inducible RNA binding protein levels in both tissues and serum.
- Healthy control group: 40 healthy controls from who skin biopsies and blood samples will be taken to assess serum and tissue levels of cold-inducible RNA binding protein and compare them to active cases.

SUMMARY:
Lichen planus (LP) is a chronic inflammatory mucocutaneous disease of unknown etiology.

Pathogenesis of LP is not completely understood, but it's considered a T-cell-mediated autoimmune disease. Cold-inducible RNA binding protein (CIRP or CIRBP) is a member of the glycine-rich RNA-binding protein family, Recent studies proved that CIRP acts as a tumor promoter through its actions on different cellular proliferation levels, Recently, the role of the damage associated molecular proteins and cytokines was highlighted in the pathogenesis of many disorders including psoriasis, alopecia areata, vitiligo, rheumatoid arthritis, other autoimmune diseases as well as several types of cancer. The aim of this study is to compare serum and tissue levels of CIRP in patients with LP and healthy controls.

DETAILED DESCRIPTION:
The aims of this study are:

* Assessment of serum and tissue levels of CIRP in patients with LP.
* To compare serum and tissue levels of CIRP in patients with LP and healthy controls.
* To compare CIRP levels according to LP severity. A cross-sectional study will be conducted on 40 patients with LP and 40 age and gender matched healthy controls. Diagnosis of LP will be clinically and will be confirmed by dermoscopy.

  * Methods of the study:

    1. Evaluation of CIRP expression:

       Every participant in this study will be subjected to both blood sampling and skin biopsy taking in the same session, then each sample will be processed separately and blindly at the Clinical Pathology, and Histology Departments as following:
* Blood sampling:

Three ml venous blood sample will be taken from every one of the two studied groups in a free anticoagulant tube, enabling the blood to be coagulated. After 30 minutes of leaving the tube at room temperature till coagulation, then samples will be centrifuged (at 3000 rpm for 15 min) and the resultant serum will be stored at -80c until testing (22). Serum CIRP levels will be measured using an enzyme-linked immunosorbent assay analysis (ELISA) kit.

• Skin biopsies: One skin biopsy will be taken with 3 mm punch from each patient and control. These biopsies will be taken under local anesthesia from LP lesions and the same areas matched in control. All biopsies will be submitted to Histology Department, Sohag Faculty of Medicine. They will be fixed in 10% neutral buffered formalin, dehydrated in ascending grades of ethanol followed by immersion in xylene then impregnated in paraffin. Several 5 micron (5um) thick sections from each block will be taken. One slide will be stained by hematoxylin and eosin (H&E) for routine histopathological examination. Other sections will be mounted on positive charged slides and stored at room temperature to be stained immunohistochemically.

1. Histopathological assessment of H&E-stained sections:

   Sections stained with H&E will be evaluated under the light microscope to confirm the diagnosis of LP and to asses epidermal and dermal changes.
2. Immunohistochemical (IHC) staining procedure The method used for immunostaining will be streptavidin-biotin amplified system. Paraffin-embedded tissue sections will be deparaffinized in xylene, rehydrated in a graded series of ethanol, and incubated with 3% hydrogen peroxide. Slides will be rinsed in phosphate - buffered saline (PBS) and then exposed to heat-induced epitope retrieval in citrate buffer solution (Ph 6) for 20 minutes. After cooling, the slides will be incubated over night at room temperature with mouse monoclonal anti-CIRP antibody (0.1 ml concentrated and diluted by PBS in a dilution 1:75). Detection of immunoreactivity will be carried out using the Universal Labeled Streptavidin-Biotin system, horseradish peroxidase. Finally, the reaction will be visualized by an appropriate substrate/ chromogen (diaminobenzidine) reagent. The staining procedure will include the negative controls obtained by substitution of primary antibodies with phosphate-buffered saline (16).
3. Interpretation of CIRP immunostaining:

The CIRP immunostaining will be assessed separately and blindly in LP lesion and control cases. Epidermal and dermal cells will be assigned positive by the presence of brownish coloration detected by DAB reaction either in the cytoplasm or nuclei in ≥ 1 stained cells (25).

ELIGIBILITY:
Inclusion Criteria:

* Patients from both sexes aged 18 - 60 years, having clinical and dermoscopic confirmed LP and did not receive any topical or systemic treatment in the last 3 months for LP.

Exclusion Criteria:

1 . Pregnancy and lactation. 2. Patients with any infections or sepsis. 3. Patients with any other dermatological diseases associated with increased CIRP levels (eg. psoriasis, vitiligo or alopecia areata).

4. Patients with systemic illness (cardiac, renal, hepatic or respiratory), malignancy, with history of connective tissue diseases or on immunosuppressive treatment.

5. Patients who received any topical or systemic treatment for LP 3 months before the study.

6. Patients with oral, nail or scalp LP.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 40 patients with LP and 40 age and gender matched healthy controls who will attend the Dermatology Outpatient Clinics, Sohag University Hospitals. Diagnosis of LP will be clinically and will be confirmed by dermoscopy.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of cold-inducible RNA binding protein levels in serum and tissue | about one year
  Skin biopsies and blood samples will be taken to assess CIRBP levels

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A Abu El-Hamd, MD, Study Chair — Sohag University; Soha H Aboeldahab, MD, Study Director — Sohag University; Rasha I Mohamed, MD, Study Director — Sohag University
Locations (1):
- Aya Ahmed Elsayed, Sohag, Egypt